CLINICAL TRIAL: NCT06140810
Title: Impact of Atelectasis and Lung Recruitment on RVEDP Measurement in Children Undergoing Cardiac Catheterization for Surveillance Following Orthotropic Heart Transplantation
Brief Title: Impact of Atelectasis on RVEDP Following Orthotropic Heart Transplantation
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Baylor College of Medicine (Other)
Responsible Party: Principal Investigator, Adam Adler MD, MS, FAAP, Associate Professor of Anesthesiology, Baylor College of Medicine
Other Study IDs: H52547
Record Dates: First submitted 2023-11-15; First posted 2023-11-20 (Actual); Last update posted 2023-12-21 (Actual); Status verified 2023-12

CONDITIONS: Heart Transplant Failure; Anesthesia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Right ventricular End diastolic pressure: Measurement of pre and post recruitment right ventricular end diastolic pressure
  Interventions: Other: Lung Recruitment

INTERVENTIONS:
Other: Lung Recruitment — Lung Recruitment will be performed during general anesthesia to reduce areas of atelectasis

SUMMARY:
Following orthoptopic heart transplantation (OHT), children undergo surveillance cardiac catheterizations to assess for signs of rejection including muscle biopsy as well as pressure measurements to guide post transplant treatment regiments. These procedures are done under general anesthesia which promotes lung tissue collapse (atelectasis). What is not known is the effect of atelectasis on intracardiac pressures which are a critical area of monitoring post-transplant patients for rejection.

DETAILED DESCRIPTION:
Following orthoptopic heart transplantation (OHT), children undergo surveillance cardiac catheterizations to assess for signs of rejection including muscle biopsy as well as pressure measurements. These procedures are done under general anesthesia which promotes lung tissue collapse (atelectasis). Atalectaisis is known to alter intra-thoracic pressures and cardiac loading conditions. What is not known is the effect of atelectasis on intracardiac pressures which are a critical area of monitoring post-transplant patients for rejection. Therefore, the aim of this study is to identify if atelectasis impacts the pressure measurements obtained during cardiac catheterization.

ELIGIBILITY:
Inclusion Criteria:

* Patients having undergone orthotropic heart transplantation
* Patients requiring routine heart catheterization for post-transplant surveillance
* General anesthesia

Exclusion Criteria:

* Patient/parental refusal
* Patients with suspected or known acute rejection
* Known anti-rejection medication non-compliance
* Patients within 1 year following heart transplant
* Home oxygen requirement
* Previous lung surgery (e.g., lobectomy) other than biopsy
* Lung transplantation
* Known pulmonary fibrosis
* Known pulmonary hypertension (>1/2 systemic)
* Sedation without the use of an airway device
* Active respiratory infection -Inability to provide recruitment breaths >25mmHg -Cardiomegaly
* Recipient/donor size mismatch

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: This is a study in patients following orthotropic heart transplantation meeting the inclusion exclusion criteria.
Sampling Method: Probability Sample
Enrollment: 15 (Estimated)
Dates: Start 2023-11-20 (Actual); Primary Completion 2024-11-01 (Estimated); Study Completion 2024-11-01 (Estimated)

PRIMARY OUTCOMES:
Number of participants with reduction of right ventricular end diastolic pressure of 3mmHg or greater | 10 minutes
  Change of the right ventricular end diastolic pressure from pre and post recruitment breaths

CONTACTS AND LOCATIONS:
Overall Officials: adam adker, MD, Principal Investigator — Texas Childrens Hospital
Locations (1):
- Texas Childrens Hospital, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: Undecided
De-identified data will be made available upon written request